CLINICAL TRIAL: NCT00116727
Title: Rheumatoid Arthritis Disease Modifying Anti-Rheumatic Drug (DMARD) Intervention and Utilization Study (RADIUS 2)
Brief Title: Rheumatoid Arthritis DMARD Intervention and UtilizationStudy
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Other Study IDs: 20021635; 016.0035
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; DMARD
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Drug: etanercept 50 mg/wk SC
  Interventions: Drug: ENBREL®

INTERVENTIONS:
Drug: ENBREL® — 50 mg/wk SC

SUMMARY:
To systematically collect and document use patterns, effectiveness and safety of DMARD treatments currently used in the management of rheumatoid arthritis. The primary purpose of this study is to estimate the incidence of serious adverse experiences and adverse experiences of interest in patients with rheumatoid arthritis (RA) treated with ENBREL®.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the 1987 American Rheumatism Association criteria for RA
* Currently requiring the addition of ENBREL® therapy (to be taken alone or in addition to their current DMARD therapy)

Exclusion Criteria:

* Currently or previously enrolled in RADIUS 1
* Currently enrolled in a clinical trial where treatments or patient visits are imposed by a protocol
* Active infections
* Known allergy to ENBREL® or any of its components
* Current treatment with ENBREL®
* Patients who have previously been demonstrated to be intolerant of or refractory to ENBREL® therapy
* Nursing or pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients (by ACR criteria) starting on etanercept alone or in combination with other DMARDs
Sampling Method: Non-Probability Sample
Enrollment: 5103 (Actual)
Dates: Start 2002-10; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Gibofsky A, Palmer WR, Keystone EC, Schiff MH, Feng J, McCroskery P, Baumgartner SW, Markenson JA. Rheumatoid arthritis disease-modifying antirheumatic drug intervention and utilization study: safety and etanercept utilization analyses from the RADIUS 1 and RADIUS 2 registries. J Rheumatol. 2011 Jan;38(1):21-8. doi: 10.3899/jrheum.100347. Epub 2010 Oct 15. PMID 20952478
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com